CLINICAL TRIAL: NCT02118129
Title: Knowledge, Attitudes, Intake and Blood Levels of Vitamin D Among Young Adults: an Intervention Study Using a Mobile 'App'.
Brief Title: Vitamin D Among Young Adults: an Intervention Study Using a Mobile 'App'.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Vitamin D Society (Other)
Responsible Party: Principal Investigator, Kelly Anne Meckling, PhD, Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014GoodmanVitD
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Intervention; Behaviour; Mobile app
MeSH Terms: conditions — Vitamin D Deficiency; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioural intervention (Experimental): Behavioural intervention consisting of an educational video component and use of a handheld mobile app to track vitamin D intake.
  Interventions: Behavioral: an educational video
- Control group (Placebo Comparator): Wait-list control group
  Interventions: Other: wait listed

INTERVENTIONS:
Behavioral: an educational video
  Arms: Behavioural intervention
Other: wait listed
  Arms: Control group

SUMMARY:
The purpose of this study is to examine whether a behavioural intervention changes attitudes, knowledge, intake or blood levels of vitamin D in young adults. The hypothesis is that an educational component and use of a mobile smartphone 'app' will increase knowledge and/or intake of vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-25 years
* Must be fluent in English
* Must be currently living in Canada
* Must own iPhone, iPad or iPod Touch running iOS 7.0 or higher (handheld 'app' used in intervention is only available in Apple Store; not available for Android or Blackberry platforms at this time)

Exclusion Criteria:

* Outside age group
* Not fluent in English
* Not living in Canada
* Does not own the specified Apple device

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Vitamin D blood levels | 12 weeks
  Blood will be collected by finger prick at baseline and after the 12-week behavioural intervention to measure 25(OH)D.
Vitamin D Intake | 12 weeks
  Vitamin D intake will be assessed using a food frequency questionnaire before and after the 12-week intervention.

SECONDARY OUTCOMES:
Knowledge & attitudes regarding vitamin D | 12 weeks
  General knowledge & attitudes regarding vitamin D will be assessed via online questionnaire before, mid-way and after the 12-week intervention.

OTHER OUTCOMES:
Vitamin D app recordings | 12 weeks
  Participants will enter their intake of foods & beverages into a handheld mobile 'app'. The data will produce a daily total intake of calcium & vitamin D. This data will be analyzed to assess changes in vitamin D intake throughout the 12-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly A Meckling, PhD, Principal Investigator — University of Guelph; Samantha E Goodman, MSc, Study Director — University of Guelph; Barbara A Morrongiello, PhD, Study Director — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goodman S, Morrongiello B, Meckling K. A randomized, controlled trial evaluating the efficacy of an online intervention targeting vitamin D intake, knowledge and status among young adults. Int J Behav Nutr Phys Act. 2016 Nov 11;13(1):116. doi: 10.1186/s12966-016-0443-1. PMID 27836017